CLINICAL TRIAL: NCT06234982
Title: Jodkids: a Study of Iodine Intake Among Children Aged 2-10 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DTU National Food Institute (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Gitte Ravn-Haren, Senior Researcher, Technical University of Denmark
Other Study IDs: DTUNationalFoodInstitute
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-01

CONDITIONS: Diet Habit; Iodine Deficiency; Iodine Toxicity
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 2-3 years of age: 2-3 years of age
- 4-6 years of age: 4-6 years of age
- 7-10 years of age: 7-10 years of age

SUMMARY:
The overall aim of the study is to monitor the effects of the increased iodine fortification level implemented in 2019 on iodine intake from the diet (incl. dietary supplements) and the excretion of iodine in urine in children aged 2-10 years.

DETAILED DESCRIPTION:
All children in Denmark receive iodine fortification through the iodine fortification program of salt, bread, and baked goods. As DANSDA's results demonstrate a risk of increased iodine intake among the youngest children, it is necessary to carry out the study in these age groups, as this can have harmful effects on children's thyroid health as well as neural development. Children are the group in society that most easily exceeds the intake of iodine, whereas many pregnant women still find it difficult to achieve a sufficient intake with the current level of fortification. Through this study, it is possible to detect and deal with a potentially too high intake in children in time. If, on the other hand, the study shows that the children have a satisfactory intake of iodine, the iodine fortification level can potentially be increased, so that the iodine intake is increased in the groups that still have an iodine intake below the recommended level.

The study consists of two sub-studies. The specific objectives of the sub-studies are to:

* Iodine status (1): Estimate the iodine intake and food sources of iodine among children after the increased iodine fortification and assess whether some children are at risk of an increased iodine intake (2-10 years old).
* Diet validation (2): Validate the estimated iodine intake based on dietary records against the actual iodine intake measured in spot urines (4-10-year-olds).

A total of 600 participants are recruited, divided into 200 participants in each of three age groups: 1) 2-3 years, 2) 4-6 years and 3) 7-10 years. A short, electronic questionnaire is completed for all participants. In the iodine status study (1), the child's parents/guardians collect one urine spot sample from each participant to measure the population's iodine intake. The diet validation study (2) is carried out in a subsample of 100 participants divided into 50 participants in each of the age groups 2) 4-6 years and 3) 7-10 years. From here, the child's parents/guardian register data for the dietary intake every day for 7 consecutive days and collect one spot urine per day on the same 7 days when the dietary registration takes place.

All examinations are considered harmless.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-10 years

Exclusion Criteria:

* Chronic diseases that can influence iodine metabolism (metabolic diseases, kidney or liver diseases or diabetes)
* Parents/guardians do not have the opportunity to fill in the basic questionnaire or the diet questionnaire electronically

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of approximately 600 children aged 2-10 years. The sample includes children in nursery, kindergarten and school up until 5th grade.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Urinary Iodine Excretion | Baseline
  Iodine and creatinine in urine samples

SECONDARY OUTCOMES:
Iodine intake | Baseline
  Dietary intake assessed by a 7-day web-based food diary
BMI | Baseline
  Weight and height will be combined to report BMI in kg/m^2
Socio-demographic background information | Baseline
  Questionnaire about parents' education

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Ravn-Haren, Ph.D, Principal Investigator — DTU National Food Institute
Locations (1):
- Technical University of Denmark, Kongens Lyngby, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No